CLINICAL TRIAL: NCT05959863
Title: LC-MS/MS-specific Cutoffs for Screening and Confirmatory Testing of Primary Aldosteronism: A Multi-center Study
Brief Title: Primary Aldosteronism LC-MS/MS-specific Cutoffs
Acronym: PM
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Collaborators: Chinese PLA General Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Qifu Li, Professor, Chongqing Medical University
Other Study IDs: PM-China 2023
Record Dates: First submitted 2023-06-26; First posted 2023-07-25 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Primary Aldosteronism
Keywords: Diagnostic; Multicenter study
MeSH Terms: conditions — Hyperaldosteronism; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Aldosteronism Group: Patients diagnosed with primary aldosteronism
  Interventions: Diagnostic Test: Captopril Challenge Test
- Essential Hypertension Group: Patients diagnosed with essential hypertension
  Interventions: Diagnostic Test: Captopril Challenge Test

INTERVENTIONS:
Diagnostic Test: Captopril Challenge Test — Patients received 50 mg captopril orally in the morning after sitting or standing for at least two hours. PAC and PRC were measured using mass spectrometry two hours after administration of capopril.

SUMMARY:
Aims to evaluation the LC-MS/MS-specific cutoffs of PA screening and CCT test.

DETAILED DESCRIPTION:
Plasma aldosterone concentration and plasma renin activity / concentration measurement are important for early screening and diagnosis of Primary Aldosteronism (PA), most measurement methods are currently based on chemiluminescence, which may be cross-reactivity with other compounds and metabolites, leading to misdiagnosis or missed diagnosis of PA patients. Liquid chromatography tandem mass spectrometry (LC-MS/MS) has been introduced into the clinical routine analysis of steroid hormones due to its higher specificity and is increasingly used for the diagnosis of adrenal diseases. However, it is unknown for the cut-offs of PA screening and CCT test based on this technology in China. Therefore, the purpose of this study is to establish the screening and CCT cut-off point for primary aldosteronism based on LC-MS/MS technique at multicenter in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age is between 18-75 years old.
2. Hypertension patients with high risk factors for PA (meeting one of the following criteria): a.Persistent hypertension (> 150 / 100mmHg); b. Refractory hypertension (combined with 3 antihypertensive drugs and one used as a diuretic,Blood pressure is still greater than 140 / 90 mmHg or four antihypertensive drugs are needed to control blood pressure of less than 140 / 90 mmHg); c.Hypertension with adrenal accidental tumor; d.Hypertension is associated with hypokalaemia;
3. Recent and stable use of antihypertensive drugs for more than 2 weeks, The drug types may include: β receptor blockers, CCB(calcium channel blockers), angiotension converting enzyme inhibitors(ACEi), Angiotensin Receptor Blocker(ARB), mineralocorticoid receptor antagonists(MRA), and other diuretics.

Exclusion Criteria:

1. Patients who are unwilling to participate and complete the study or refuse to sign a written informed consent for the study;
2. Patients diagnosed with other secondary hypertension (such as renal hypertension, renal artery stenosis, pheochromocytoma, Cushing's syndrome, etc.);
3. Combined with severe renal insufficiency eGFR <30 ml/min / 1.73 m2, Or patients with liver insufficiency OR liver failure (Alanine aminotransferase and / or aspartate aminotransferase increased 2.5 times above the upper limit of normal);
4. Clinical assessment of a dressing change risk, Including: Heart failure (NYHA stage grade II or above), any one or more of the stroke, myocardial infarction, and unstable angina pectoris diagnosed within three months;
5. Patients who are pregnant or who are currently being treated with sex hormones and glucocorticoids;
6. incurable malignancy;
7. Other reasons make it difficult to change or stop the drug to complete the diagnosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study intends to include patients taking hypertension medication at each center between June 2023 and July 2024 with subjects signing written informed consent.
Sampling Method: Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Establish a LC-MS/MS assay-specific cut-off point of screening without medication interfering for primary aldosteronism. | At baseline without medication interfering.
  Measure the plasma aldosterone concentration and plasma renin activity by LC-MS/MS.Plasma aldosterone concentration and plasma renin activity will be combined and reported as an aldosterone-to-renin ratio.
Establish a LC-MS/MS assay-specific cut-off point of CCT without medication interfering for primary aldosteronism. | 2 hours after the captopril challenge test without medication interfering.
  Measure the plasma aldosterone concentration by LC-MS/MS.

SECONDARY OUTCOMES:
Establish a LC-MS/MS assay-specific cut-off point of screening with medication interfering for primary aldosteronism. | At baseline with medication interfering.
  Measure the plasma aldosterone concentration and plasma renin activity by LC-MS/MS.
  Plasma aldosterone concentration and plasma renin activity will be combined and reported as an aldosterone-to-renin ratio.
compare the different criteria of Captopril Challenge Test for the diagnosis of primary aldosteronism. | 2 hours after the captopril challenge test without medication interfering.
  plasma aldosterone concentration were measured using automated chemiluminescence immunoassays.

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (2):
- China (2):
  - Qifu Li, Chongqing, Chongqing Municipality
  - Department of Endocrinology, the First Affiliated Hospital of Chongqing Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulatero P, di Cella SM, Monticone S, Schiavone D, Manzo M, Mengozzi G, Rabbia F, Terzolo M, Gomez-Sanchez EP, Gomez-Sanchez CE, Veglio F. 18-hydroxycorticosterone, 18-hydroxycortisol, and 18-oxocortisol in the diagnosis of primary aldosteronism and its subtypes. J Clin Endocrinol Metab. 2012 Mar;97(3):881-9. doi: 10.1210/jc.2011-2384. Epub 2012 Jan 11. PMID 22238407
- [Result] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Result] Fuss CT, Brohm K, Kurlbaum M, Hannemann A, Kendl S, Fassnacht M, Deutschbein T, Hahner S, Kroiss M. Confirmatory testing of primary aldosteronism with saline infusion test and LC-MS/MS. Eur J Endocrinol. 2021 Jan;184(1):167-178. doi: 10.1530/EJE-20-0073. PMID 33112272
- [Result] Young WF Jr. Diagnosis and treatment of primary aldosteronism: practical clinical perspectives. J Intern Med. 2019 Feb;285(2):126-148. doi: 10.1111/joim.12831. Epub 2018 Sep 25. PMID 30255616
- [Result] Olsen MH, Angell SY, Asma S, Boutouyrie P, Burger D, Chirinos JA, Damasceno A, Delles C, Gimenez-Roqueplo AP, Hering D, Lopez-Jaramillo P, Martinez F, Perkovic V, Rietzschel ER, Schillaci G, Schutte AE, Scuteri A, Sharman JE, Wachtell K, Wang JG. A call to action and a lifecourse strategy to address the global burden of raised blood pressure on current and future generations: the Lancet Commission on hypertension. Lancet. 2016 Nov 26;388(10060):2665-2712. doi: 10.1016/S0140-6736(16)31134-5. Epub 2016 Sep 23. No abstract available. PMID 27671667
- [Result] Rehan M, Raizman JE, Cavalier E, Don-Wauchope AC, Holmes DT. Laboratory challenges in primary aldosteronism screening and diagnosis. Clin Biochem. 2015 Apr;48(6):377-87. doi: 10.1016/j.clinbiochem.2015.01.003. Epub 2015 Jan 22. PMID 25619896